CLINICAL TRIAL: NCT05251662
Title: A Phase II Study of Sintilimab Combined With GEMOX ± IBI305 (Bevacizumab Biosimilar) Versus GEMOX as First-line Therapy in Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Sintilimab Combined With GEMOX ± IBI305 (Bevacizumab Biosimilar) Versus GEMOX in Advanced Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGBICC
Record Dates: First submitted 2022-01-11; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; First-line Therapy; Sintilimab; IBI305; GEMOX
MeSH Terms: conditions — Cholangiocarcinoma | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group1 (Experimental): Sintilimab Combined With GEMOX + IBI305
  Interventions: Drug: Sintilimab; Drug: IBI305; Drug: GEMOX
- experimental group2 (Experimental): Sintilimab Combined With GEMOX
  Interventions: Drug: Sintilimab; Drug: GEMOX
- Comparator (Active Comparator): GEMOX
  Interventions: Drug: GEMOX

INTERVENTIONS:
Drug: Sintilimab — 200mg IV d1 Q3W
  Arms: experimental group1; experimental group2
Drug: IBI305 — 7.5mg/kg IV d1 Q3W
  Other Names: Bevacizumab Biosimilar
  Arms: experimental group1
Drug: GEMOX — Oxaliplatin 100mg/m2 IV d1 Q3W+ gemcitabine 1000mg/m2 IV d1/8 Q3W

SUMMARY:
A randomized controlled, phase II clinical trial is designed to compare the safety and efficacy of Sintilimab combined with GEMOX ± IBI305 and GEMOX as first-line therapy in advanced intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent should be signed before implementing any trial-related procedures
* Male or female, 18 years old ≤ age ≤ 75 years old
* Histopathologically or cytologically diagnosed as locally advanced intrahepatic cholangiocarcinoma
* No previous systemic treatment, More than 6 months after the end of postoperative adjuvant therapy was allowed
* Expected survival time > 3 months
* At least ≥ 1 measurable lesions per RECIST 1.1
* ECOG PS scores 0-2
* Sufficient organ and bone marrow function
* Urine or serum pregnancy test is negative

Exclusion Criteria:

* Suffered from other malignant tumors in the past 5 years (except Radical basal cell carcinoma of the skin squamous carcinoma of the skin and/or radical resected carcinoma in situ)
* Ampullary tumor
* Received treatment from other clinical trials within 4 weeks before the first dose
* Received any anti-PD-1 antibody, anti-PD-L1/L2 antibody, anti-CTLA4 antibody, or other immunotherapy
* Suffered from severe cardiovascular disease within 12 months before enrollment, such as symptomatic coronary heart disease, congestive heart failure ≥ Grade II, uncontrolled arrhythmia, and myocardial infarction
* Uncontrollable pleural effusion, pericardial effusion or ascites
* Use steroids or other systemic immunosuppressive therapies 4 weeks before enrollment
* Allergic reactions to the drugs used in this study
* HIV antibody positive, active hepatitis B or C (HBV, HCV)
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* other conditions that the investigator deems inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2025-01-13 (Estimated)

PRIMARY OUTCOMES:
Overall response rate ( ORR) | up to 90 days after last treatment administration
  Overall response rate ( ORR) is defined as proportion of participants who have a best response of CR or PR

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 90 days after last treatment administration
  Disease Control Rate (DCR) is defined as proportion of participants who have a best response of CR、PR or SD
Progression free survival (PFS) | up to 3 years
  the time period from randomization of the participants to objective tumor progression or death
Overall survival (OS) | up to 3 years
  the time period from the randomization of the participants to the death event due to any reason
Adverse event | up to 30 days after last treatment administration
  All grades of adverse events, all grades of treatment related adverse events, serious of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China